CLINICAL TRIAL: NCT04083521
Title: The Effect of Bacillus Subtilis DE111® on the Daily Bowel Movement Profile for People With Occasional Gastrointestinal Irregularity
Brief Title: Effect of Bacillus Subtilis DE111® on Daily Bowel Movements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deerland Enzymes (Industry)
Collaborators: Kennesaw State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DE111Reg
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Bowel Movement Regulation; Occasional Constipation; Occasional Diarrhea
Keywords: Bowel movement regulation; Occasional constipation; Occasional diarrhea; Gastrointestinal health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Subjects received a once daily dose of Bacillus subtilis DE111® 1x10^9 CFU for 90-days.
  Interventions: Dietary Supplement: Bacillus subtilis DE111®
- Placebo (No Intervention): Subjects received a once daily dose of maltodextrin for 90-days.

INTERVENTIONS:
Dietary Supplement: Bacillus subtilis DE111® — Subjects were administered a dose of Bacillus subtilis at levels of 1x10^9 CFU once a day for 90-days.
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine the efficacy of Bacillus subtilis DE111® probiotic for regulation of bowel movements.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy of the probiotic B. subtilis DE111® for regulation of bowel movements. A single capsule containing 1 x 10^9 CFU B. subtilis is to be consumed once a day per participant. 50 adults (18-65 years of age at the time of participation) suffering from occasional constipation and/or diarrhea will be enrolled. Participants will be double-blindly and randomly assigned to either the probiotic (Bacillus subtilis) or the placebo (maltodextrin) group. Efficacy will be assessed with participant-reported bowel movement (BM) records. As a secondary outcome, the study will provide further insight into the tolerance of the supplement. Tolerance will be assessed using a digestive health questionnaire and blood samples to analyze pertinent metabolic biomarkers. Participants will be asked to complete a daily dietary intake record as well. Prior to capsule consumption, participants will complete a two-week pre-testing phase in order to provide a more inclusive diagnostic baseline. This phase will consist of daily BM and dietary intake record keeping.

ELIGIBILITY:
Inclusion Criteria:

* Participants suffering from occasional constipation and/or diarrhea will be eligible for participation.

Exclusion Criteria:

* Blood CRP levels for each participant will be monitored at days 0, 60 and 105 of this study. Participants with CRP levels greater than 5mg/l on day 0 of the study will be excluded from further participation as this level is indicative of underlying inflammatory bowel disease. Participants excluded under such conditions will be instructed to seek further treatment with their health care provider.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Bowel movement regularity | 105-day study period (consisting of 90-days treatment plus 15-day follow up)
  Increasing regularity of bowel movements in subjects with occasional diarrhea or constipation
Tolerance | 105-day study period (consisting of 90-days treatment plus 15-day follow up)
  To determine if the supplement is tolerable among subjects without causing adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: No